CLINICAL TRIAL: NCT04659967
Title: Hearing Loss and Communication Needs in a Group Care Setting for Older Adults
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Massachusetts, Amherst (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Principal Investigator, Sara Mamo, Assistant Professor, University of Massachusetts, Amherst
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 680; 1K23DC016855 (NIH)
Record Dates: First submitted 2020-12-02; First posted 2020-12-09 (Actual); Last update posted 2022-05-06 (Actual); Status verified 2022-05

CONDITIONS: Age-related Hearing Loss
MeSH Terms: conditions — Presbycusis

STUDY DESIGN:
Intervention Model Description: Staff will be invited to participate in an experiential virtual sensitivity training. A pre/post quasi-experimental design will be undertaken. Staff will be asked to complete a pre-training questionnaire as well as follow-up questionnaires immediately after the training and one month, three months, and six months post training to measure knowledge gained and to probe for behavior change related to the communication strategies taught during the training. Some participants who complete questionnaires will be contacted and invited to participate in a research interview about their communication experiences at PACE. The training session will last for up to 1 hour. All questionnaires are expected to take approximately 15 minutes each. Interviews will take 1-hour.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pre/Post Training (Within subject) (Experimental): Participants will complete a baseline questionnaire followed by immediate virtual training, and complete a post-training questionnaire. Participants will also be asked to complete a questionnaire 1-month, 3-months, and 6-months post-training.
  Interventions: Behavioral: Virtual Training

INTERVENTIONS:
Behavioral: Virtual Training — Participants will receive a virtual training that is tailored to age-related hearing loss, use of non-custom personal amplification devices, and communication strategies.

SUMMARY:
The purpose of this study is to develop and test a multicomponent hearing care intervention for the PACE staff members in order to learn more about communication and engagement.

DETAILED DESCRIPTION:
The long-term objective of this proposal is to increase the accessibility and affordability of hearing loss treatment for older adults with hearing loss, with a particular interest in adults that have mild cognitive impairment (MCI) or dementia. Age-related hearing loss (ARHL) in persons with MCI or dementia may exacerbate dementia-related symptoms such as depression, apathy, agitation/aggression. Moreover, engagement and activity participation are recognized as critical aspects of dementia care management, but those individuals who also experience ARHL are at a disadvantage. A pilot testing of behavioral communication intervention will be completed at multiple Program for All-inclusive Care for the Elderly (PACE) sites in New England. A multicomponent hearing care intervention will be tested that includes staff training and non-custom personal amplification use with older adults in a group care setting. This feasibility study will lead to the refinement of the intervention protocols to be used in a future grant application that will test the real-world efficacy of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* PACE staff who work in the Day Health Center and are available to attend the training on-site at PACE are eligible for inclusion. All staff are invited to join the training (via Zoom, if necessary), but to complete the research activities, they have to complete the training in-person due to the hands-on component of learning to use the hearing device.

Exclusion Criteria:

* Staff members who cannot attend the (virtual) in-person training.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-12-02 (Actual); Primary Completion 2021-11-22 (Actual); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline on a Hearing communication Knowledge Assessment at 1 Month. | 1 month follow-up
  Participants will complete a questionnaire to monitor retention of communication strategies and behaviors.
Change From Baseline on a Hearing communication Knowledge Assessment at 3 Months. | 3 month follow-up
  Participants will complete a questionnaire to monitor retention of communication strategies and behaviors.
Change From Baseline on a Hearing communication Knowledge Assessment at 6 Months. | 6 month follow-up
  Participants will complete a questionnaire to monitor retention of communication strategies and behaviors.

SECONDARY OUTCOMES:
Qualitative Interviews | 6-12 months post training
  We will purposefully sample staff members whose quantitative results indicate that they were either successful or unsuccessful in learning and using new communication behaviors.

CONTACTS AND LOCATIONS:
Overall Officials: Sara K Mamo, AuD, PhD, Principal Investigator — University of Massachusetts, Amherst
Locations (3):
- United States (3):
  - PACE Upham's Elder Service Plan, Boston, Massachusetts
  - Mercy LIFE PACE, West Springfield, Massachusetts
  - PACE Organization of Rhode Island, Providence, Rhode Island

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ciorba A, Bianchini C, Pelucchi S, Pastore A. The impact of hearing loss on the quality of life of elderly adults. Clin Interv Aging. 2012;7:159-63. doi: 10.2147/CIA.S26059. Epub 2012 Jun 15. PMID 22791988
- [Background] Chen DS, Betz J, Yaffe K, Ayonayon HN, Kritchevsky S, Martin KR, Harris TB, Purchase-Helzner E, Satterfield S, Xue QL, Pratt S, Simonsick EM, Lin FR; Health ABC study. Association of hearing impairment with declines in physical functioning and the risk of disability in older adults. J Gerontol A Biol Sci Med Sci. 2015 May;70(5):654-61. doi: 10.1093/gerona/glu207. Epub 2014 Dec 3. PMID 25477427
- [Background] Cohen-Mansfield J, Taylor JW. Hearing aid use in nursing homes. Part 1: Prevalence rates of hearing impairment and hearing aid use. J Am Med Dir Assoc. 2004 Sep-Oct;5(5):283-8. PMID 15357885
- [Background] Genther DJ, Betz J, Pratt S, Kritchevsky SB, Martin KR, Harris TB, Helzner E, Satterfield S, Xue QL, Yaffe K, Simonsick EM, Lin FR; Health ABC Study. Association of hearing impairment and mortality in older adults. J Gerontol A Biol Sci Med Sci. 2015 Jan;70(1):85-90. doi: 10.1093/gerona/glu094. Epub 2014 Jul 14. PMID 25024235
- [Background] Genther DJ, Betz J, Pratt S, Martin KR, Harris TB, Satterfield S, Bauer DC, Newman AB, Simonsick EM, Lin FR; Health, Aging and Body Composition Study. Association Between Hearing Impairment and Risk of Hospitalization in Older Adults. J Am Geriatr Soc. 2015 Jun;63(6):1146-52. doi: 10.1111/jgs.13456. Epub 2015 Jun 11. PMID 26096388
- [Background] Haque, R., Abdelrehman, N., & Alavi, Z. (2012). "There's a monster under my bed": Hearing aids and dementia in long-term care settings. Annals of Long-Term Care, 20(8), 28-33.
- [Background] Hopper, T., & Hinton, P. (2012). Hearing loss among individuals with dementia: Barriers and facilitators to care. Canadian Journal of Speech-Language Pathology & Audiology, 36(4), 302-313.
- [Background] Hopper TL. "They're just going to get worse anyway": perspectives on rehabilitation for nursing home residents with dementia. J Commun Disord. 2003 Sep-Oct;36(5):345-59. doi: 10.1016/s0021-9924(03)00050-9. PMID 12927943
- [Background] Lin FR, Albert M. Hearing loss and dementia - who is listening? Aging Ment Health. 2014;18(6):671-3. doi: 10.1080/13607863.2014.915924. No abstract available. PMID 24875093
- [Background] Lin FR, Metter EJ, O'Brien RJ, Resnick SM, Zonderman AB, Ferrucci L. Hearing loss and incident dementia. Arch Neurol. 2011 Feb;68(2):214-20. doi: 10.1001/archneurol.2010.362. PMID 21320988
- [Background] Lin FR, Yaffe K, Xia J, Xue QL, Harris TB, Purchase-Helzner E, Satterfield S, Ayonayon HN, Ferrucci L, Simonsick EM; Health ABC Study Group. Hearing loss and cognitive decline in older adults. JAMA Intern Med. 2013 Feb 25;173(4):293-9. doi: 10.1001/jamainternmed.2013.1868. PMID 23337978
- [Background] Mamo SK, Nirmalasari O, Nieman CL, McNabney MK, Simpson A, Oh ES, Lin FR. Hearing Care Intervention for Persons with Dementia: A Pilot Study. Am J Geriatr Psychiatry. 2017 Jan;25(1):91-101. doi: 10.1016/j.jagp.2016.08.019. Epub 2016 Sep 22. PMID 27890543
- [Background] Mick P, Kawachi I, Lin FR. The association between hearing loss and social isolation in older adults. Otolaryngol Head Neck Surg. 2014 Mar;150(3):378-84. doi: 10.1177/0194599813518021. Epub 2014 Jan 2. PMID 24384545
- [Background] Lin FR, Hazzard WR, Blazer DG. Priorities for Improving Hearing Health Care for Adults: A Report From the National Academies of Sciences, Engineering, and Medicine. JAMA. 2016 Aug 23-30;316(8):819-20. doi: 10.1001/jama.2016.7916. No abstract available. PMID 27254725
- [Background] Nieman CL, Marrone N, Mamo SK, Betz J, Choi JS, Contrera KJ, Thorpe RJ Jr, Gitlin LN, Tanner EK, Han HR, Szanton SL, Lin FR. The Baltimore HEARS Pilot Study: An Affordable, Accessible, Community-Delivered Hearing Care Intervention. Gerontologist. 2017 Nov 10;57(6):1173-1186. doi: 10.1093/geront/gnw153. PMID 27927734